CLINICAL TRIAL: NCT00523562
Title: Study of the Role of Insulin Resistance in the Pathogenesis of the Metabolic Syndrome and of Non-alcoholic Steatohepatitis
Brief Title: Effects of Macronutrients on Hepatic Lipids, Plasma Triglycerides, and Insulin Sensitivity
Acronym: MACRONUTR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Responsible Party: Principal Investigator, Luc Tappy, MD, Professor Luc Tappy, University of Lausanne
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: protocol 140/04/CE/FBM
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Metabolic Syndrome X; Liver Diseases
Keywords: fructose; dietary lipids; dietary proteins; hepatic steatosis; insulin resistance; Healthy humans; overweight humans; obese humans
MeSH Terms: conditions — Metabolic Syndrome; Liver Diseases; Fatty Liver; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- normal weight male high fructose diet (Experimental): Effects of diet intervention " high fructose" in normal weight subjects
  Interventions: Other: diet intervention
- offsprings of T2DM high fructose diet (Experimental): Effect of diet intervention "high fructose" in healthy non-obese offsprings of patients with type 2 diabetes
  Interventions: Other: diet intervention
- normal weight subjects high fat diet (Experimental): effects of diet intervention "high fat" in healthy male subjects
  Interventions: Other: diet intervention
- Normal weight high fat+protein diet (Experimental): effect of diet intervention "high fat + protein" subjects in healthy male subjects
  Interventions: Other: diet intervention

INTERVENTIONS:
Other: diet intervention — controlled hypercaloric high fructose, high fat, or high fat/high protein diet

SUMMARY:
The purpose of this study is to assess how the macronutrient composition of the diet effects

* lipid and glucose metabolism
* intrahepatic lipids
* insulin sensitivity

in healthy lean subjects and in subjects with a high metabolic risk (ie overweight and offsprings of patients with type 2 diabetes mellitus).

DETAILED DESCRIPTION:
The study is aimed at assessing the effects of changes in total energy, sugars, lipids, and protein intake on intrahepatic lipids, plasma lipids, and hepatic and whole body insulin resistance in

* lean men and women with no family history of diabetes
* overweight men and women
* lean men with a family history of type 2 diabetes

Subjects are studied after a 6-day period of

* isocaloric diet with 100% calorie requirement, of which 55% carbohydrate, 15% protein, and 30% fat)
* the same isocaloric diet supplemented with 3g/kg body weight/day fructose
* hypercaloric high fat diet with 130% energy requirement, of which 55% carbohydrate, 15% protein, 60% fat
* hypercaloric high fat+protein diet with 145% energy requirement, of which 55% carbohydrate, 30% protein, 60% fat

Measurements performed after 6 days on each diet include

* intrahepatic and intramyocellular lipids (1H-MRS)
* hepatic and whole body insulin sensitivity (hyperinsulinemic-euglycemic clamp)
* body weight
* plasma concentrations of hormones and substrates
* gene expression profile in skeletal muscle (vastus lateralis) and adipose tissue (subcutaneous abdominal)

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age 18-40
* Informed consent obtained
* Subgroup with overweight (body mass index [BMI] > 25)
* Subgroup with family history of type 2 diabetes mellitus

Exclusion Criteria:

* Smokers
* Alcohol intake > 30g/day
* Drug abuse
* Diabetes mellitus
* Any concurrent medication
* Having a pacemaker
* History of orthopedic surgery
* History of metal foreign bodies

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2006-07; Primary Completion 2008-04 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
plasma triglycerides | 6 days
intra-hepatic lipids | 6 days
insulin mediated glucose disposal | 6 days

SECONDARY OUTCOMES:
lipid oxidation | 6 days
plasma beta-hydroxybutyrate | 6 days
gene expression in skeletal muscle and adipose tissue | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Luc Tappy, MD, Principal Investigator — University of Lausanne
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

REFERENCES:
- [Derived] Bortolotti M, Kreis R, Debard C, Cariou B, Faeh D, Chetiveaux M, Ith M, Vermathen P, Stefanoni N, Le KA, Schneiter P, Krempf M, Vidal H, Boesch C, Tappy L. High protein intake reduces intrahepatocellular lipid deposition in humans. Am J Clin Nutr. 2009 Oct;90(4):1002-10. doi: 10.3945/ajcn.2008.27296. Epub 2009 Aug 26. PMID 19710199
- [Derived] Le KA, Ith M, Kreis R, Faeh D, Bortolotti M, Tran C, Boesch C, Tappy L. Fructose overconsumption causes dyslipidemia and ectopic lipid deposition in healthy subjects with and without a family history of type 2 diabetes. Am J Clin Nutr. 2009 Jun;89(6):1760-5. doi: 10.3945/ajcn.2008.27336. Epub 2009 Apr 29. PMID 19403641